CLINICAL TRIAL: NCT00002572
Title: Intracavitary Allogenic Cytotoxic T Lymphocytes and Human Recombinant Interleukin-2 Therapy for Recurrent Primary Brain Tumors
Brief Title: Cytotoxic T Cells and Interleukin-2 in Treating Adult Patients With Recurrent Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 93-0426.cc; UCHSC-COMIRB-93426; NCI-T94-0065O
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2000-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Gliosarcoma | interventions — aldesleukin; Muromonab-CD3

INTERVENTIONS:
Biological: aldesleukin
Biological: muromonab-CD3
Biological: therapeutic tumor infiltrating lymphocytes
Procedure: conventional surgery

SUMMARY:
RATIONALE: Biological therapy uses different ways to stimulate the immune system and stop cancer cells from growing. Cytotoxic T cells combined with interleukin-2 may be an effective treatment for recurrent brain tumors.

PURPOSE: Phase I trial to study the effectiveness of cytotoxic T cells and interleukin-2 in treating adults with recurrent brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the toxicity of allogeneic cytotoxic T lymphocytes (CTL) when repeatedly instilled directly into the brain to treat recurrent primary brain tumors. II. Evaluate the response produced by allogeneic CTL and interleukin-2. III. Correlate CTL surface phenotype and degree of patient/donor HLA mismatch to response and toxicity.

OUTLINE: Surgery plus Biological Response Modifier Therapy. Tumor resection; plus intracavitary cytotoxic T lymphocytes, CTL; intracavitary Interleukin-2 (Chiron), IL-2, NSC-373364. CTL are generated in vitro by mixing irradiated patient lymphocytes (cultured with IL-2 and Monoclonal Antibody OKT 3, MOAB OKT 3, NSC-618843) with allogeneic lymphocytes and culturing the mixture with IL-2.

PROJECTED ACCRUAL: 10 patients will be treated. If severe toxicity occurs in the first 5 patients, the study will close.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Kernohan Grade III/IV primary malignant brain tumor that has failed conventional surgical resection and radiotherapy Evidence of recurrent tumor on gadolinium-enhanced MRI following completion of radiotherapy (minimum 5,000 cGy for adults) required The following histologies are eligible: Anaplastic astrocytoma Anaplastic oligodendroglioma Glioblastoma multiforme Mixed anaplastic glioma Surgical resection of progressing brain tumor feasible No evidence of tumor extending across the midline from one hemisphere to the other No multifocal tumor or leptomeningeal spread

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Karnofsky 60-100% Life expectancy: At least 2 months Hematopoietic: WBC greater than 2,000 Platelets greater than 100,000 Hct at least 28% Hepatic: Bilirubin less than 1.5 mg/dl Renal: Creatinine less than 1.5 mg/dl Cardiovascular: No major cardiovascular problems Pulmonary: No major pulmonary problems Other: Seronegative for HTLV/HIV, syphilis, and hepatitis B and C No concurrent systemic infection Ability to maintain proper nutrition (orally or intravenously) during the study period required No pregnant women

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: More than 4 weeks since systemic chemotherapy (6 weeks since carmustine), with the WBC increasing on 2 consecutive determinations at least 3 days apart Endocrine therapy: Not specified Radiotherapy: At least 8 weeks since radiotherapy Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 1994-11; Primary Completion 1999-12 (Actual); Study Completion 1999-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin O. Lillehei, MD, Study Chair — University of Colorado, Denver
Locations (3):
- United States (3):
  - Children's Health Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado